CLINICAL TRIAL: NCT00635323
Title: A Phase 2 Study of the Efficacy and Safety of Irinotecan (Campto®) in Combination With Capecitabine (Xeloda®) as First-Line Chemotherapy in Asian Subjects With Inoperable Hepatocellular Carcinoma
Brief Title: Safety And Efficacy Of Irinotecan Plus Capecitabine As First-Line Treatment In Asian Subjects With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP4174/2501; A5961080
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Irinotecan plus capecitabine

INTERVENTIONS:
Drug: Irinotecan plus capecitabine — Irinotecan 200-250 mg/m2 intravenous infusion over 30 to 90 minutes on day 1 of a 3-week cycle. Capecitabine 1000 mg/m2 oral tablet twice daily for 14 days followed by a 7 day rest throughout the treatment period for

SUMMARY:
To evaluate the safety and efficacy of irinotecan and capecitabine in Asian subjects with inoperable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Asian subjects with histologically or cytologically confirmed hepatocellular carcinoma
* Inoperable disease (unable to completely remove surgically, presence of extra-hepatic disease, main portal vein or hepatic vein involvement)
* Eastern Cooperative Oncology Group performance status of ?2

Exclusion Criteria:

* Decompensated cirrhosis or stage C (Index>10) according to the Child-Pugh Classification
* Current history of chronic diarrhoea
* Reproductive potential not using adequate contraceptive measures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2002-11; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Week 6

SECONDARY OUTCOMES:
Time to progression | Weeks 6, 12, 18, 24, 36, and 1 year
Duration of overall response | Weeks 6, 12, 18, 24, 36, and 1 year
Overall tumour growth control rate | Weeks 6, 12, 18, 24, 36, and 1 year
Overall survival | Weeks 6, 12, 18, 24, 36, and 1 year
Adverse events | Weeks 6, 12, 18, 24, 36, and 1 year
Physical exam | Weeks 6, 12, 18, 24, 36, and 1 year
Laboratory tests | Weeks 6, 12, 18, 24, 36, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Pfizer Investigational Site, Shanghai, China
- Pfizer Investigational Site, Hong Kong SAR, Hong Kong
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (2):
  - Pfizer Investigational Site, Keelung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XRP4174/2501&StudyName=Safety%20And%20Efficacy%20Of%20Irinotecan%20Plus%20Capecitabine%20As%20First-Line%20Treatment%20In%20Asian%20Subjects%20With%20Hepatocellular%20Carcinoma